CLINICAL TRIAL: NCT01642901
Title: Zoledronic Acid to Prevent Bone Loss After Acute Spinal Cord Injury
Brief Title: Zoledronic Acid in Acute Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11F.612
Record Dates: First submitted 2012-07-06; First posted 2012-07-17 (Estimated); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; bone mineral density
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Zoledronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic Acid 5 mg IV infusion (Experimental): Single infusion of 5 mg intravenous zoledronic acid given within 21 days of acute traumatic spinal cord injury.
  Interventions: Drug: Zoledronic acid
- normal saline 0.9% (Placebo Comparator): Infusion of normal saline of equivalent volume to reconstituted zoledronic acid, given only once and run over 2 hours, to occur within 21 days of acute traumatic spinal cord injury.
  Interventions: Drug: normal saline 0.9%

INTERVENTIONS:
Drug: Zoledronic acid — 5 mg zoledronic acid infused intravenously over two hours (2.5mg per hour), given only once, within 21 days of acute traumatic spinal cord injury.
  Other Names: Reclast
  Arms: Zoledronic Acid 5 mg IV infusion
Drug: normal saline 0.9% — Infusion of equivalent volume of 0.9% normal saline to that of the reconstituted zoledronic acid, given only once over two hours, occurring within 21 days of acute traumatic spinal cord injury
  Other Names: normal saline; 0.9% saline
  Arms: normal saline 0.9%

SUMMARY:
Maintenance of bone mass following spinal cord injury (SCI) is essential to fracture prevention and the associated morbidity of bed rest and further secondary complications. Intravenous (IV) zoledronic acid (ZA) is an FDA-approved drug that has been shown to be more effective than other agents in reducing bone mass resorption and leg fractures in post-menopausal women, but has not been studied in patients with acute SCI. This will be a randomized, double-blind, placebo-controlled trial of IV ZA to prevent bone loss early after SCI. Up to 48 subjects will be randomized to receive a one-time dose of 5 mg of IV ZA versus placebo within 21 days of an SCI.

DETAILED DESCRIPTION:
Maintenance of bone mass following spinal cord injury (SCI) is essential to fracture prevention and the associated morbidity of bed rest and further secondary complications. Intravenous (IV) zoledronic acid (ZA) has been shown to be more effective than other agents in reducing bone mass resorption and fracture of the legs in post-menopausal women, but has not been studied in acute spinal cord injury. Two previous studies of ZA in persons with subacute SCI, while promising, were inconclusive. As stated in the long range plan of the National Institute on Disability and Rehabilitation Research (NIDRR), one goal in the area of health and function is to "focus on the onset of new conditions…exacerbation of existing conditions, or the development of coexisting conditions." This study is intended to demonstrate reduction in loss of bone mass at the hip and knee regions in acute SCI in a rigorous study of sufficient size to determine effectiveness of our intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65, male or female
* Traumatic SCI with Neurological level C4-T10, American Spinal Injury Association (ASIA) Impairment Scale (AIS) A,
* Serum calcium level >7.0 mg/dL) at time of study drug administration
* Screening baseline serum 25-hydroxy (25-OH) vitamin D of at least 13 ng/ml
* No medical contraindication to supplemental vitamin D for participants whose levels are >13 ng/ml but sub-therapeutic (<32ng/ml)
* No medical contraindication to supplemental calcium
* Weight under 300 pounds, which is the maximum permitted on the dual-energy X-ray absorptiometry (DXA) scanner

Exclusion Criteria:

* Ventilator-dependent individuals
* Chronic steroid use (defined as >6 months)
* Rheumatoid disease with use of prior disease modifying anti-rheumatic drugs (DMARDs) affecting bone density
* History of osteoporosis or of treatment for osteopenia or osteoporosis with bisphosphonates, or selective reuptake estrogen modifying agents
* Current use of medications* including bisphosphonates to treat osteoporosis (*note that prior calcium or vitamin D use is not an exclusion criteria)
* History of more than one lower extremity osteoporosis-related fracture
* Chronic renal insufficiency, creatinine clearance < 35 ml/min, during screening
* End stage liver or kidney disease
* Medical conditions resulting in hypogonadal states that affect bone density
* Uncontrolled thyroid disease/thyrotoxicosis
* Hereditary or acquired metabolic bone disorder
* History of use of unfractionated heparin for >1 year
* History of selected antiseizure medications, specifically phenobarbital, phenytoin, carbamazepine, sodium valproate >1 year
* Acute or chronic bilateral lower extremity fractures involving tibia or femur, with placement of surgical hardware in any areas of above locations
* Severe hypotension requiring use of intravenous blood pressure agents such as dopamine, norepinephrine or phenylephrine. Exception may allow for patients on pressors who arm experiencing hypotension as they acclimate to upright posture.
* Inability to provide informed consent and understand the consent process
* Facial fractures requiring oral surgery
* Dental surgery or oral maxillofacial surgery within 2 weeks of anticipated study drug administration
* Pregnancy present on admission
* Vitamin D deficiency on admission testing (serum 25-OH D reported as < 13 ng/mL)
* Patients with an established reaction to, or history of, anaphylactic shock to aspirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina V Oleson, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University and Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oleson CV, Marino RJ, Formal CS, Modlesky CM, Leiby BE. The effect of zoledronic acid on attenuation of bone loss at the hip and knee following acute traumatic spinal cord injury: a randomized-controlled study. Spinal Cord. 2020 Aug;58(8):921-929. doi: 10.1038/s41393-020-0431-9. Epub 2020 Feb 13. PMID 32055041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two comprehensive acute inpatient rehabilitation facilities between September 2012 and March 2017.
Pre-assignment Details: Prior to day 10 post injury, investigators obtained serum calcium, intact parathyroid hormone and serum 25-hydroxy (25-OH) vitamin D levels to determine further eligibility. Participants with vitamin D deficiency were allowed to receive supplementation to raise their level above 13 ng/mL in order to participate. One participant who was consented was subsequently found to have facial fractures and was withdrawn prior to randomization.
Period: Intervention
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Started | 10 | 5
Completed | 10 (One participant had knee flexion contractures and spasticity that prevented accurate DXA at the knee.) | 5
Not Completed | 0 | 0
Period: 4-month Follow-up
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0
Period: 12-month Follow-up
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Started | 10 | 5
Completed | 9 (One participant had knee flexion contractures and spasticity that prevented accurate DXA at the knee.) | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9% | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (12.6) | 30.8 (9.9) | 34.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 3 | 9
  Black | 2 | 2 | 4
  Hispanic | 1 | 0 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15
Total proximal femur areal bone mineral density (aBMD) [Mean (Standard Deviation); unit: g/cm^2] | 0.98 (0.076) | 1.09 (0.138) | 1.02 (0.108)
Intertrochanteric femur aBMD [Mean (Standard Deviation); unit: g/cm^2] | 1.15 (0.094) | 1.28 (0.147) | 1.19 (0.126)
Femoral neck aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.86 (0.078) | 0.98 (0.178) | 0.90 (0.127)
Distal femur aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.88 (0.092) | 1.01 (0.128) | 0.924 (0.118)
Proximal tibia aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.94 (0.138) | 1.11 (0.217) | 1.00 (0.180)
serum C-telopeptide (CTX) [Mean (Standard Deviation); unit: pg/ml] | 1255 (704) | 980 (439) | 1163 (626)
procollagen N-1 terminal propeptide (P1NP) [Mean (Standard Deviation); unit: mcg/L] | 67.9 (37.9) | 52.8 (9.50) | 62.9 (31.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Areal Bone Mineral Density at Hip
Description: Percent change in areal bone mineral density (aBMD) assessed by dual energy X-ray absorptiometry (DXA) at 4 months compared to baseline.
  This will compare aBMD at the hip.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 10 | 5
percentage change
  Total proximal femur | 0.92 (7.14) | -12.0 (7.50)
  Intertrochanteric femur | 1.19 (7.77) | -12.9 (7.67)
  Femoral neck | 0.97 (6.12) | -9.37 (6.39)

2. Primary Outcome: Change in Areal Bone Mineral Density at Knee
Description: Percent change in areal bone mineral density (aBMD) assessed by dual energy X-ray absorptiometry (DXA) at 4 months compared to baseline.
  This will compare aBMD at the distal femur and proximal tibia.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 9 | 5
percentage change
  Distal femur | -0.78 (4.46) | -6.75 (4.04)
  Proximal tibia | -0.24 (11.7) | -8.56 (14.1)

3. Primary Outcome: Change in Areal Bone Mineral Density at Hip
Description: Percent change in areal bone mineral density (aBMD) assessed by dual energy X-ray absorptiometry (DXA) at 12 months post-injury compared to baseline.
  This will compare aBMD at the hip.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 10 | 5
percentage change
  Total proximal femur | -8.2 (3.64) | -21.3 (8.66)
  Intertrochanteric femur | -8.62 (4.70) | -19.4 (7.00)
  Femoral neck | -3.93 (5.60) | -17.0 (11.8)

4. Primary Outcome: Change in Areal Bone Mineral Density at Knee
Description: Percent change in areal bone mineral density (aBMD) assessed by dual energy X-ray absorptiometry (DXA) at 12 months post-injury compared to baseline.
  This will compare aBMD at the distal femur and proximal tibia.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 8 | 5
percentage change
  Distal femur | -8.07 (5.2) | -10.0 (8.7)
  Proximal tibia | -4.54 (9.89) | -10.0 (18.3)

5. Secondary Outcome: Change in Biomarkers of Bone Resorption (sCTX)
Description: Change in sCTX from baseline to 1- and 4-months post intervention and 12-months post-injury.
Time Frame: 1 month, 4 months, 12 months
Population: Ons subject in each group did not return for 12-month labs
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 10 | 5
percentage change
  1 month | -64.1 [-73.4 to -60.8] | 14.4 [11.5 to 15.5]
  4 months | -45.9 [-51.4 to -25.6] | 23.9 [-11.9 to 62.3]
  12 months: number analyzed (Participants) | 9 | 4
  12 months | -43.6 [-57.9 to 33.5] | -5.11 [-38.2 to 10.9]

6. Secondary Outcome: Change in Biomarkers of Bone Formation (P1NP)
Description: Change in serum P1NP from baseline to 1- and 4-months post intervention.
Time Frame: 1 month, 4 months
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 10 | 5
percentage change
  1 month | 5.66 [-1.19 to 54.05] | 65.96 [48.08 to 101.96]
  4 months | 32.43 [3.70 to 113.21] | 27.45 [18.84 to 213.33]

7. Secondary Outcome: Safety and Tolerability of Zoledronic Acid
Description: Assessment of the safety and tolerability of zoledronic acid in the acute spinal cord injury population. This will be done by examination reportable adverse events including fevers, flu-like symptoms, GI upset as measures of safety and report of patient's willingness to have participate in physical therapy in the first week after receiving medication as a measure of tolerability
Time Frame: 72-hours and 1 month post intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
Number analyzed (Participants) | 10 | 5
Participants
  Fever > 100.9 within 72 hours of study drug infusion | 7 | 1
  Flu-like symptoms within 72 hours of study drug infusion | 6 | 1
  Acute kidney injury | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 month
Description: Subject #7 developed chest pain within 24-hours of study drug administration. Cardiac workup was negative but laboratory studies found elevated creatine phosphokinase (CPK). Baseline and periodic serum CPK studies over the first 7 days after study drug administration were added to the protocol for subsequent patients.
Arm/Group | Zoledronic Acid 5 mg IV Infusion | Normal Saline 0.9%
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/5
Other Adverse Events (participants affected / at risk) | 7/10 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid 5 mg IV Infusion (N=10) | Normal Saline 0.9% (N=5)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Zoledronic Acid 5 mg IV Infusion (N=10) | Normal Saline 0.9% (N=5)
Fever (General disorders) | 7 (7) | 1 (1) — Temperature greater than or equal to 101 degrees Fahrenheit within 72 hours of study drug administration
Flu-like symptoms (General disorders) | 6 (6) | 1 (1) — Flu-like symptoms within 72 hours of study drug administration
elevated creatine phosphokinase (CPK) (Musculoskeletal and connective tissue disorders) | 1/6 (1) | 0/3 (0)

LIMITATIONS AND CAVEATS:
Enrollment was significantly less than projected due to competing acute clinical trials, reducing the power of the study to identify significant differences.

DXA imaging, particularly at the knee was limited by positioning on the table in some individuals with evolving contractures in either knee flexion or hip rotation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT01642901/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT01642901/ICF_001.pdf